CLINICAL TRIAL: NCT02760446
Title: Validation of the French Confusion Assessment Method for the Intensive Care Unit Among Adult ICU Patient
Brief Title: Translation and Validation of the French Version of Confusion Assessment Method for the Intensive Care Unit
Acronym: CAM-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9596
Record Dates: First submitted 2015-12-22; First posted 2016-05-03 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Patients With Mental Confusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAM-ICU.fr (Other): CAM-ICU and ICDSC evaluation proceed by two investigators and a Neuropsychologist (Speech & language therapist specialized in neuropsychology)
  Interventions: Behavioral: CAM-ICU.fr

INTERVENTIONS:
Behavioral: CAM-ICU.fr — Neuropsychological testing

SUMMARY:
Validity and Reliability of French Version of the Confusion Assessment Method for the Intensive Care Unit (psychometric validation study after translation/back translation process assessed by the original team : W.Ely, MD, Ph.D, Vanderbilt University)

ELIGIBILITY:
Inclusion Criteria:

* Adult, > or equal to 18-yr
* Richmond Agitation Sedation Scale (RASS) > or equal -3
* Francophone

Exclusion Criteria:

* Diagnostic of cognitive disorders
* Admission for brain injury
* Psychotic disorders
* Diagnostic of cognitive disorders
* Visual or auditory impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Statistical criteria of performance (sensibility, specificity, negative predictive value, positive predictive value) of Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) compared to gold standard (neuropsychologist). | Day 0
  Investigators team: evaluation by the CAM- ICU in French and Intensive Care Delirium Screening Check list (ICDSC) during 2 minutes for the concomitant CAM- ICU and ICDSC , carried out at 30 minutes intervals by two Clinical Research Nurse of the investigative team .
  The neuropsychologist will do the evaluation according to criteria common DSM5. Neuropsychologists now used DSM 5 criteria to diagnose delirium at our institution since new DSM 5 criteria have been published in French.

SECONDARY OUTCOMES:
Inter-rater reliability, comparison to Intensive Care Delirium Screening Checklist and standard bedside practices | Day 0
  Statistics ICDSC criteria will be assessed against the Gold Standard . The reproducibility of the CAM- ICU and ICDSC will be evaluated according to different inter-observer.

CONTACTS AND LOCATIONS:
Overall Officials: GERALD CHANQUES, MD,Ph.D, Principal Investigator — University of Montpellier Hospitals
Locations (1):
- Centre Hospitalier Universitaire Montpellier, Saint Eloi, Montpellier, Languedoc-Roussillon, France

IPD SHARING:
Plan to Share IPD: Undecided